CLINICAL TRIAL: NCT07141173
Title: Effect of Early Lifestyle Intervention on Perinatal Outcomes in High-risk Women for Gestational Hyperglycemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Central Hospital of Gynecology Obstetrics (Other)
Responsible Party: Principal Investigator, Chen Xu, Professor, Tianjin Central Hospital of Gynecology Obstetrics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025KY107
Record Dates: First submitted 2025-08-18; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: GDM
Keywords: GDM; RCT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Individual lifestyle management
  Interventions: Behavioral: Individual lifestyle management
- control group (No Intervention): control group

INTERVENTIONS:
Behavioral: Individual lifestyle management — Manage the diet, exercise, weight and healthy lifestyle of pregnant women
  Arms: Intervention Group

SUMMARY:
This study aims to explore whether early intervention for high-risk groups of gestational hyperglycemia can improve insulin resistance and effectively prevent the occurrence of GDM, and evaluate which pathophysiological subtypes of GDM have the best effect on improving maternal and fetal adverse prognosis, so as to provide evidence for stratified management and individualized clinical intervention of high glucose groups in pregnancy

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* 6-14 weeks of pregnancy
* at least one risk factor for GDM
* signed a written informed consent

Exclusion Criteria:

* Individuals diagnosed with diabetes or prediabetes prior to pregnancy
* currently taking medications affecting blood glucose levels such as metformin
* women at risk of miscarriage
* individuals with chronic conditions (such as uncontrolled hypertension, severe heart disease)
* those with movement disorders or contraindicated conditions for physical activity
* patients undergoing gastrointestinal surgeries that alter glucose absorption
* those unable to maintain regular prenatal care (such as non-compliance with medical instructions or mental health issues).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 604 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of gestational diabetes(GDM) | 24-28 weeks pregnant
  The 75g 2h oral glucose tolerance test is performed at 24-28 weeks of gestation, and the cut-off points of venous blood glucose values are 5.1mmol/L (fasting), 10.0mmol/L (1h after glucose load), 8.5mmol/L (2h after glucose load). If any one of the three blood glucose measures is above the cut-off points, then GDM is diagnosed..

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Central Hospital of Gynecology Obstetrics, Tianjin, China

IPD SHARING:
Plan to Share IPD: No